CLINICAL TRIAL: NCT06501963
Title: Revealing Protective Immunity to Influenza Using Systems Immunology
Acronym: PRISM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Daniel S. Graciaa, MD, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00007610
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Influenza
Keywords: Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Live Attenuated Influenza Vaccine (Experimental): Participants receiving a single dose of the live attenuated influenza vaccine (LAIV).
  Interventions: Biological: Live Attenuated Influenza Vaccine

INTERVENTIONS:
Biological: Live Attenuated Influenza Vaccine — The FDA-approved live attenuated seasonal influenza vaccine (LAIV) (FluMist®, AstraZeneca) is licensed in the US for people 2-49 years of age. The approved seasonal LAIV at the time of study enrollment will be obtained from the manufacturer. LAIV will be administered by a study nurse or health care provider at the Hope Clinic as a single 0.2 milliliter (mL) dose given as 0.1 mL spray in each nostril.
  Other Names: FluMist

SUMMARY:
The goals of this study are to better understand the human immune response to influenza vaccines, specifically the live attenuated (weakened) influenza vaccine given as a nasal spray. Better understanding why this vaccine does not work as well in adults as it does in children may help design better influenza vaccines.

DETAILED DESCRIPTION:
Influenza (flu) viruses cause significant disease and death every year. Influenza vaccines protect against illness but their effectiveness can be limited. The influenza virus is notorious for its continuous mutation and potential to cause pandemics. This essentially creates a moving target for vaccine development, posing a significant challenge for global health. Current vaccines offer a certain degree of protection but are not fully effective due to the virus's ever-changing nature. In response to this, a live attenuated influenza vaccine (LAIV) was developed with the objective of providing a higher degree of protection. This type of vaccine has demonstrated remarkable effectiveness in children, surpassing the protection provided by inactivated flu vaccines. This made LAIV a preferred choice for administration to young children.

However, when it comes to adults (individuals over 18 years of age), the scenario is markedly different. Recent studies have indicated a significant decline in LAIV's effectiveness in adults compared to children. Various clinical trials have reported that LAIV exhibits approximately 85% efficacy in children under the age of 18, which dramatically decreases to around 40%-60% in adults (aged 18-49 years). This suggests that adults do not respond as well to LAIV as children do. In adults, the LAIV-induced immunity appears to be short-lived, often lasting for only one influenza season, while in children LAIV has shown to provide long-lasting protection even against mismatched strains. Understanding the factors behind this discrepancy is critical to improve the protective efficacy of influenza vaccines across all age brackets. Unraveling this mystery could open the doors to the development of a superior flu vaccine, one that offers robust protection across all age groups.

This study will enroll healthy adult (age 18-49) participants who have not received the influenza vaccine recently. Participants will be asked to come in for 3 visits over 1 month. Participants will receive the FDA-approved live attenuated influenza vaccine, given as a nasal spray. Study staff will collect baseline and follow-up biologic samples to compare how the immune system reacts. The biologic samples will be collected from the blood and nose to look at immune cells in these parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent
* Participants of child bearing potential must agree to use effective birth control for the duration of the study. A negative urine pregnancy test must be documented prior to vaccination.

Exclusion Criteria:

* History of allergy or serious adverse reaction, including Guillain-Barré syndrome, to a vaccine or vaccine products
* History of a medical condition resulting in impaired immunity such as active solid tumors, leukemia, lymphoma, chemotherapy or radiation therapy, autoimmune conditions, or splenic dysfunction. Persons with previous skin cancers or cured non-lymphatic tumors are not excluded from the study.
* History of asthma, cochlear implant, or active cerebrospinal fluid leak
* Use of immune modifying drugs including: systemic steroids for more than 1 week (such as prednisone > 20mg/day), chronic administration (more than 14 days total) of immunosuppressive or immunomodulatory drugs in the prior 3 months
* History of HIV, Hepatitis B or Hepatitis C infection
* Chronic clinically significant medical problems that could be considered active or unstable (i.e diagnosed within the past 3 months or requiring a change in medication within the past 3 months). This is including (but not limited to):

  * Insulin dependent diabetes
  * Severe heart disease (including arrhythmias)
  * Severe lung disease
  * Severe liver disease
  * Severe kidney disease
  * Severe hypertension: defined as life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit).
  * Congenital genetic syndromes (e.g., trisomy 21)
* Body Mass Index (BMI) > 35
* Pregnancy or breast feeding, or plans to become pregnant in the next month
* History of influenza infection or vaccination within the current or previous influenza season
* Receipt of blood products or immune globulin product within the prior 3 months
* History of excessive alcohol consumption, drug use, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the trial
* Receipt of any live vaccines 30 days before, or plans to receive any live vaccines 30 days after vaccination
* Receipt of any inactivated vaccines 14 days before, or plans to receive any inactivated vaccines 14 days after vaccination
* Receipt of any non-registered or other investigational product in 30 days before, or plans to receive any other investigational product 30 days after vaccination
* Temporary Exclusion Criteria:

  * Fever (temperature ≥38.0°C) or coryzal symptoms within 72 hours prior to vaccination
  * Receipt of antipyretics within 6 hours prior to vaccination

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Quantification of Antibody Titers | Day 30
  The immunogenicity of the live attenuated influenza vaccine (LAIV) is evaluated by the quantification of antibody titers using hemagglutination inhibition (HAI) assays.

SECONDARY OUTCOMES:
Mean geometric fold rise in HAI titers | Day 30
  The effect of LAIV on eliciting influenza-specific immune responses is analyzed as the mean geometric fold rise in HAI titers.
Frequency of Serious Adverse Events | Up to Day 30
  The safety profile of LAIV is assessed as the frequency of serious adverse events occurring up to 30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Graciaa, MD, MPH, MSc, Principal Investigator — Emory University
Locations (1):
- Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified immunologic assay results will be made available for sharing with other researchers.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing following publication of the results from this study.
Access Criteria: Data will be available for sharing with any researchers who wishes to access the database, or any purpose. Data will be shared via Immport (https://immport.niaid.nih.gov/home) and Zenodo (https://zenodo.org/)